CLINICAL TRIAL: NCT05193617
Title: Penpulimab Combined With GP ± Arotinib Induction Therapy + Concurrent Chemoradiotherapy + Adjuvant Peramprizumab in Locoregionally Advanced Nasopharyngeal Carcinoma: A Phase II Clinical Trial
Brief Title: Penpulimab Combined With GP ± Anlotinib as Neoadjuvant Therapy in Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Ph.D, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-FXY-504
Record Dates: First submitted 2022-01-11; First posted 2022-01-18 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP combine with Penpulimab and anlotinib neoadjuvant therapy+CCRT+Penpulimab adjuvant therapy (Experimental): Patients receive neoadjuvant therapy with gemcitabine(1000mg per square meter on days 1,8) , cisplatin (80mg per square meter on day 1), penpulimab (200mg, day1), and anlotinib (10mg days 1-14) every three weeks for three cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100mg per square meter) concurrent every three weeks during radiotherapy (D1, D22, D43 of RT) ,then followed by adjuvant therapy with penpulimab (200mg) every three weeks for a maximum of nine cycles after radiotherapy.
  Interventions: Drug: GP+Penpulimab+Anlotinib
- GP combine with Penpulimab neoadjuvant therapy+CCRT+Penpulimab adjuvant therapy (Active Comparator): Patients receive neoadjuvant therapy with gemcitabine(1000mg per square meter on days 1,8) , cisplatin (80mg per square meter on day 1), penpulimab (200mg, day1) every three weeks for three cycles before radiotherapy, then followed by concurrent IMRT and cisplatin (100mg per square meter) concurrent every three weeks during radiotherapy (D1, D22, D43 of RT) ,then followed by adjuvant therapy with penpulimab (200mg) every three weeks for a maximum of nine cycles after radiotherapy.
  Interventions: Drug: GP+Penpulimab

INTERVENTIONS:
Drug: GP+Penpulimab+Anlotinib — GP combine with penpulimab and anlotinib neoadjuvant therapy+CCRT+penpulimab adjuvant therapy
  Other Names: GP+AK105+AL3818
  Arms: GP combine with Penpulimab and anlotinib neoadjuvant therapy+CCRT+Penpulimab adjuvant therapy
Drug: GP+Penpulimab — GP combine with penpulimab neoadjuvant therapy+CCRT+penpulimab adjuvant therapy
  Other Names: GP+AK105
  Arms: GP combine with Penpulimab neoadjuvant therapy+CCRT+Penpulimab adjuvant therapy

SUMMARY:
The purpose of this study is to explore the efficacy and safety of a combination of GP chemotherapy and Penpulimab ± Anlotinib in neoadjuvant therapy combined with Penpulimab in adjuvant therapy of locoregionally advanced nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
Radiotherapy combined with chemotherapy is the standard treatment method for locally advanced NPC. In the 2020 National Comprehensive Cancer Network (NCCN) guidelines, GP regimen induction chemotherapy combined with concurrent chemoradiotherapy has been established as evidence-based grade 2A.

Based on the results of phase 3 clinical trials, the addition of PD-1 monoclonal antibody to GP chemotherapy as a first-line treatment for patients with recurrent or metastatic nonkeratinizing NPC provided superior PFS, ORR and DoR than GP alone while maintaining a manageable safety profile. Therefore, the combination of PD-1 monoclonal antibody in GP induction chemotherapy may further improve the prognosis of patients with locally advanced NPC.

There is a complex interaction between tumor immune microenvironment and tumor vascular remodeling. Anti-PD-1 monoclonal antibody combined with anti-VEGF have synergistic effect and inhibit tumor growth.

Penpulimab is a new type of PD-1 monoclonal antibody. It has the characteristics of strong antigen binding and slow dissociation rate, which can maintain the antitumor activity of T cells.

Anlotinib is a multi-target tyrosine kinase inhibitor (TKI). It can effectively inhibit a variety of receptors, including vascular endothelial growth factor receptor (VEGFR), and block tumor angiogenesis more comprehensively.

Based on the above research background, this study adopts a two-stage design:

Stage I (Pick the Winner Study): For patients with locally advanced NPC, the complete response rate (CR) of tumor after induction chemotherapy was compared between the two groups of patients receiving GP + Penpulimab and GP + Penpulimab + arotinib before radiotherapy. The regimen with higher CR rate was the winner at this stage.

Stage II ( Cohort Expansion Study): The 3-year failure free survival (FFS) of patients in the winning regimen of expansion cohort was calculated through long-term follow-up and compared with the data in previous trials.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with Written informed consent.
2. Age ≥ 18 years and ≤ 65 years, male or non-pregnant female.
3. Histologically confirmed with Nonkeratinizing carcinoma of the nasopharynx (differentiated or undifferentiated type, WHO II or III).
4. Original clinical staged as III-IVa (according to the 8th AJCC edition),exclude T3-4N0, T3N1(Only retropharyngeal lymph nodes metastasized), Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
5. White blood cell count (WBC)≥4.0×109 /L, Hemoglobin ≥ 90g/L, Platelet count ≥100×109/L.
6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN),serum total bilirubin (TBIL) ≤2.0 times the upper limit of normal (ULN) .
7. Adequate renal function: creatinine clearance rate≥60 ml/min or Creatinine ≤1.5× upper limit of normal value.

Exclusion Criteria:

1. Patients with recurrent or metastatic nasopharyngeal carcinoma.
2. Histologically or cytologically confirmed with keratinizing squamous cell carcinoma of the nasopharynx.
3. Prior therapy with Systemic chemotherapy.
4. Women in the period of pregnancy, lactation, or reproductive without effective contraceptive measures.
5. Seropositivity for human immunodeficiency virus (HIV).
6. Known history of other malignancies (except cured basal cell carcinoma or carcinoma in situ of the cervix).
7. Prior exposure to immune checkpoint inhibitors,including anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies.
8. Patients with immunodeficiency disease or a history of organ transplantation.
9. Received large doses of glucocorticoids, anticancer monoclonal antibodies, or other immunosuppressants within 4 weeks.
10. Patients with severe dysfunction of heart, liver, lung, kidney or marrow.
11. Patients with severe, uncontrolled disease or infections.
12. Received other research drugs or in other clinical trials at the same time.
13. Refuse or fail to sign the informed consent .
14. Patients with other treatment contraindications.
15. Patients with personality or mental disorders, incapacity or limited capacity for civil conduct.
16. Hepatitis B surface antigen (HBsAg) positive and peripheral blood HBV deoxyribonucleic acid (HBV DNA) ≥1000cps/ml.
17. Patients with positive HCV antibody test will only be enrolled in this study if the PCR test for HCV RNA is negative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Stage 1(Pick the Winner Study): Complete Response | 9 weeks
  The proportion of patients who had a complete response was defined as those with all pathological cervical lymph nodes being less than 10 mm in the short axis and no unequivocal soft tissue mass in the local region. Disease response was evaluatedby by the Investigator using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) 95% confidence intervals (CIs) were calculated using the Clopper Pearson method
Stage 2 (Cohort Expansion Study): Failure-free survival (FFS) | 3 years
  Defined as the time from registration to documented local or regional relapse, distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  Defined as the time from registration to death from any cause or censored at the date of last follow-up.
Locoregional failure-free survival (LRRFS) | 3 years
  Defined as the time from registration to local or regional relapse, or death from any cause.
Distant metastasis-free survival (DMFS) | 3 years
  Defined as the time from registration to distant metastasis, or death from any cause.
Incidence rate of adverse events (AEs) | 3 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) and late radiation toxicities were assessed by CTCAE v5.0.
Objective Response Rate (ORR) | 9 weeks
  Objective response rate (ORR) was assessed by the site Investigator using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1) and was defined as the percentage of patients with a confirmed overall response of complete response (CR) or partial response (PR) and was based on all treated patients who had measurable disease at baseline (Day 1). 95% confidence intervals (CIs) were calculated using the Clopper Pearson method.

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Qiang Mai, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Hai Qiang Mai, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi YR, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Liu Z, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Feng H, Yao S, Keegan P, Xu RH. Toripalimab or placebo plus chemotherapy as first-line treatment in advanced nasopharyngeal carcinoma: a multicenter randomized phase 3 trial. Nat Med. 2021 Sep;27(9):1536-1543. doi: 10.1038/s41591-021-01444-0. Epub 2021 Aug 2. PMID 34341578